CLINICAL TRIAL: NCT03867565
Title: The Role of Nutrition After Minor Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FOU2018-0249
Record Dates: First submitted 2019-01-17; First posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Burns; Nutritional Deficiency
Keywords: Minor burns; Nutrition
MeSH Terms: conditions — Burns; Malnutrition

STUDY DESIGN:
Intervention Model Description: Patients found to have nutritional diagnosis will be given tailorized nutritional intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No nutritional diagnosis (No Intervention): Patients without nutritional diagnosis get SOC
- Nutritional diagnosis (Experimental): Patients with nutritional diagnosis get nutritional intervention by dietitian.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — Indirect calorimetry Weight development Nitrogen balance Food records Physical activity Nutritional risk screening and assessment Inflammatory response Wound healing as number of days from burn to no more need of dressing changes via health care facility Frequency of infections as the number, sort, dose, and length of antibiotic treatment(s) from burn to no more need of dressing changes via health care facility
  Arms: Nutritional diagnosis

SUMMARY:
Nutrition therapy has an important role in burn care to optimize wound healing, prevent muscle wasting, improve immune function and decrease risk of infection and sepsis. The body of literature concerning major burns´nutritional requirements has increased over the last decades, however the role of nutrition after minor burns (TBSA < 20 %) is virtually unexplored and in need of further investigation. Hence, this study explores if adequate nutritional status after minor burn results in better outcome.

DETAILED DESCRIPTION:
Phase 1 Aim To study energy- and protein requirements after minor burns in adults (TBSA < 20 %).

Research questions Do energy- and protein requirements increase after minor burns? Do energy- and protein requirements proportionally increase with the severity of injury; depth and extent after minor burns? Study design/methods Sample size: 84 patients and 84 healthy control subjects (matched by age, gender and BMI).

Method: All consecutive burns, admitted for treatment at Uppsala Burn Center, fulfilling inclusion and exclusion criteria are asked to take part in this phase. Oral and written informed consent is collected. Patients background data (severity of burn injury, including depth and extent, and the treatment thereof, concomitant diseases and medications, age, weight, height, gender, socioeconomic status, alcohol- and tobacco use, physical activity level using activity meters, as well as data from questionnaire obtained from routine standard of care at Burn Center about sleep, quality of life, pain and depression) will be collected. Measure (indirect calorimetry) and calculate energy requirement (Mifflin St Jeor equation x Injury Factor x physical activity level) within 2 weeks after injury and 1, 3, 6, and 12 months after injury. Measure nitrogen balance (nitrogen balance = nitrogen intake - nitrogen loss). Collecting data from blood sample to measure inflammatory response (albumin, transferrin, CRP), if the body can use more protein (urea) and measurement of normal kidney function (cystatin-C).Collecting data from 24-h-urine collection, urea for calculation of nitrogen balance to distinguish between protein intake compared and muscle breakdown. Data for calculation of protein intake from nutritional assessment and 4-day food record. Results are compared with 84 healthy control subjects measured with indirect calorimetry, blood sample, urine collection, and intake measurement.

Phase 2 Aim To describe nutritional status in adult patients after minor burns. Nutritional status is defined as to what degree physiological nutrient needs are met (energy- and protein intake compared to measurements and calculations, carbohydrate-, fat-, vitamin-, and mineral intake compared to estimated average requirements. Weight and muscle mass compared to normal body composition and its development over time).

Research questions Do minor burns affect nutritional status? Does nutritional status differ related to injury severity? Sample size: 84 patients included in Phase 1 are asked to take part in this study.

Method: All consecutive burns, admitted for treatment at the Uppsala Burn Center, fulfilling inclusion and exclusion criteria are asked to take part in this phase. Oral and written informed consent is collected. Patients background data from phase 1 will be collected.

Screening for nutritional risk, identifying mild, moderate and severe impaired nutritional status (undernourishment): screening tool, NRS 2002 (19), within 2 weeks from injury, and follow-up 1, 3, 6, and 12 months after injury. Screening is performed by a dietitian.

Nutritional assessment: data from phase 1 will be collected about intake, energy- and protein needs, weight and muscle mass. Dietary history interview, to collect data about patients' intake the year before injury.

Nutritional diagnosis of malnutrition (16) were nutritional risk screening and nutritional assessment will provide the basis for diagnosis.

Phase 3 Aim To identify types of nutritional diagnoses, and nutritional interventions, and the effects on signs and symptoms for respective nutritional diagnosis, in adults after minor burns.

To create a nutrition algorithm for nutritional interventions after minor burns.

Research questions Frequency of different types of aetiologies to identify nutritional diagnoses? Frequency of different types of nutritional diagnoses? Frequency and types of nutritional interventions? Is the nutrition diagnosis treated by the nutrition intervention (fully, partly, not)? Results of nutritional interventions (variable depends on signs and symptoms relevant for respective nutritional diagnosis e.g. energy- and protein intake)? Study design/methods Sample size: Patients identified as in need of nutritional intervention in phase 2 are asked to take part in this study.

Method: Oral and written informed consent is collected. Patients background data from phase 1 will be collected.

Nutritional intervention: Nutritional intervention is initiated with follow-up at dietitian's discretion. Nutrition Care Process is used:

1. Assessing patient data (material from phases 1-2 and additional assessment at dietitian's discretion)
2. Diagnosing nutritional problems (for example inadequate protein- energy intake, inadequate protein intake, food- and nutrition- knowledge deficit, unintended weight loss, malnutrition) and determining the problems´ aetiologies
3. Implementing one or more interventions (for example recommendations on meal frequency, foodstuff, use of nutritional support, education on basics)
4. Monitoring and evaluating patient progress (compliance to nutritional interventions, and sign and symptoms relevant for respective nutritional diagnosis, e.g. weight change, energy- and protein intake) Compliance to nutritional interventions: evaluated by assessing patient data at follow-up (asking patients about compliance to treatment during nutritional assessment).

Weight development: Weekly the patients' weight will be measured as long as patients have a nutritional treatment. Thereafter at follow-up 1, 3, 6, and 12 months after injury. During the patients´ stay/visits at the burn center this is done at the hospital. Thereafter to no more need of dressing changes via health care facility patients will measure weight at home/external health facility and report the number to the clinic.

Phase 4 Aim To study the role, in adults, of nutrition after minor burns (TBSA < 20 %) on outcome (wound healing and infections and body weight).

Research questions Do nutritional status and food/supplement intake affect time to heal wounds, frequency of infections, and weight changes, after minor burns? Study design/methods Sample size: 84 patients included in phase 1 are asked to take part in this phase.

Method:

All consecutive burns, admitted for treatment at the Uppsala Burn Center, fulfilling inclusion and exclusion criteria are asked to take part in the study. Oral and written informed consent is collected. Patients background data from phase 1 will be collected.

Wound healing: As surrogate parameter for number of days to wound healing the number of days from burn to no more need of dressing changes via health care facility will be measured. During routine clinical visits to the burn center, photography of wounds will be taken. Three blinded plastic surgeons with burn care experience will assess the photos for % of initial wound healed correlated to days from burn.

Frequency of infections: As surrogate parameter for frequency of infections the number, sort, dose, and length of antibiotic treatment(s) during the period from burn to no more need of dressing changes via health care facility will be measured.

Weight development: Weekly the patients´ weight will be measured. During the patients´ stay/visits at the burn center this is done at the hospital. Thereafter to no more need of dressing changes via health care facility patients will measure weight at home/external health facility and report the number to the clinic.

Nutritional assessment: Data from phases 1, 2 and 3, energy- and protein requirements, nutritional intake, muscle mass and nutritional diagnoses and the treatment thereof.

ELIGIBILITY:
Inclusion Criteria:

* Minor burn, TBSA < 20 %
* Age ≥ 18 years old
* Understands Swedish or English verbally and in writing
* Mentally adequate
* Oral and written informed consent.

Exclusion Criteria:

* Patients deemed not to be able to complete study protocol.
* TBSA < 2 %.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2023-03-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Change in energy balance from trauma to 12 months after minor burns | within 2 weeks after injury, 1, 3, 6, 12 month after injury
  Resting energy expenditure (REE) measured by indirect calorimetry to study energy requirements. REE are added with measurement of physical activity level (PAL) from 4-day activity measurement and compared to energy intake (that are collected from 4-day food record) to analyze energy balance.
Change in nitrogen intake from trauma to 12 months after minor burns | Measured within 2 weeks after injury, 1, 3, 6, 12 months after injury.
  Nitrogen intake is measured and calculated from a 4-day food record
Change in nitrogen loss from trauma to 12 months after minor burns | Measured within 2 weeks after injury, 1, 3, 6, 12 months after injury.
  Nitrogen loss is calculated from 24-h-urine collection (urea).
Weight development from trauma to 12 months after minor burns | Every week after trauma until no more need for dressing changes via health care facility and also within 2 weeks after injury, 1, 3, 6, 12 months after injury.
  Weight will be measured every week after trauma until no more need for dressing changes via health care facility. For all patients´ weight will also be measured within 2 weeks after injury, 1, 3, 6, 12 months after injury. During the patients´ stay/visits at the burn center this is done at the hospital. Thereafter weight will be measured at home/external health facility.
Frequency of infection from trauma to 12 months after minor burns | within 2 weeks after injury, 1, 3, 6, 12 month after injury
  As surrogate parameter for frequency of infections the number, sort, dose, and length of antibiotic treatment(s) during the period
Wound healing from trauma to 12 months after minor burns | Every week after trauma until no more need for dressing changes via health care facility and also within 2 weeks after injury, 1, 3, 6, 12 months after injury
  As surrogate parameter for number of days to wound healing the number of days from burn to no more need of dressing changes via health care facility will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik RM Huss, Ass Prof, Principal Investigator — Burn Center, Dept. of Plastic and Maxillofacial Surgery

IPD SHARING:
Plan to Share IPD: No